CLINICAL TRIAL: NCT07123662
Title: A Clinical Study on the Safety and Efficacy of γδ T Cells in Preventing Relapse After Allogeneic Transplantation in High-risk Acute Myeloid Leukemia Patients
Brief Title: γδ T Cell Therapy for Relapse Prevention in High-Risk AML Post-Transplant
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-24-021
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Leukemia; Myeloid; Acute
Keywords: γδ T cells; AML; Prevent recurrence
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamma-Delta T cell injection (Experimental): Experimental group: Received γδT infusion after high-risk AML allogene transplantation standard prophylactic treatment.
  Interventions: Biological: Gamma-Delta T cell injection
- Standard prophylactic treatment (Other): Control group: High-risk AML received only standard prophylactic treatment after allogeneic transplantation
  Interventions: Other: Standard prophylactic treatment

INTERVENTIONS:
Biological: Gamma-Delta T cell injection — Experimental group: Peripheral intravenous infusion of γδ T cells
  Arms: Gamma-Delta T cell injection
Other: Standard prophylactic treatment — Standard prophylactic treatment
  Arms: Standard prophylactic treatment

SUMMARY:
This is a prospective, double-arm, single-center, randomized controlled single-blind clinical study

DETAILED DESCRIPTION:
This study is a prospective, single-center, two-arm, single-blind randomized controlled clinical trial to evaluate the safety and efficacy of γδ T cell infusion in preventing recurrence in patients with high-risk AML after allogeneic transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily sign informed consent and are expected to complete the follow-up examination and treatment of the study procedures;
2. Age 18-65 years old (including cut-off value), gender is not limited;
3. AML patients have one of the high-risk factors for recurrence after allogeneic hematopoietic stem cell transplantation;
4. AML patients need to meet 30±5 days after the end of allogeneic transplant therapy;
5. The patient has recovered from the toxicity of the prior treatment, i.e., CTCAE toxicity grade < 2 (unless the abnormality is related to the tumor or is stable as judged by the investigator and has little impact on safety or efficacy);
6. ECOG performance status score of 0-3 points and expected survival greater than 3 months ;
7. Have appropriate organ function:

   1. Alanine aminotransferase (ALT) ≤3 times the upper limit of normal (ULN);
   2. Aspartate aminotransferase (AST) ≤ 3 times ULN;
   3. Total bilirubin ≤1.5 times ULN;
   4. Serum creatinine ≤1.5 times ULN or creatinine clearance ≥ 60 mL/min;
   5. Hemoglobin ≥ 50g/L (must not have received transfusion support within 7 days prior to laboratory tests);
   6. Room oxygen saturation ≥92%;
   7. Left ventricular ejection fraction (LVEF) ≥ 45%, echocardiography confirmed no pericardial effusion, no clinically significant ECG findings;
   8. Without clinically significant pleural effusion;

Exclusion Criteria:

1. Other malignant tumors within 3 years prior to screening, except for adequately treated carcinoma in situ of the cervix, papillary carcinoma of the thyroid, basal cell or squamous epithelial cell skin cancer, localized prostate cancer after radical resection, and ductal carcinoma in situ after radical resection;
2. Patients have a severe allergic history;
3. The patient has severe heart disease;
4. The patient has severe respiratory system disease;
5. Those with grade III~IV acute GVHD or extensive chronic GVHD;
6. Patients who are using (or willing to use) other maintenance therapy drugs after hematopoietic stem cell transplantation and have proven that this maintenance therapy drug is not conducive to the persistence of γδ T cells in vivo;
7. Active neurological autoimmune or inflammatory diseases, amyotrophic lateral sclerosis (ALS), and clinically significant active cerebrovascular disease;
8. Patients with severe mental illness;
9. Alcoholics or those with a history of drug abuse;
10. Clinically significant active cerebrovascular disease;
11. Those who have participated in other clinical studies within 1 month before screening and have not interfered with the safety and efficacy of this study drug as assessed by the investigator are allowed to be included in the study, such as non-interventional observational studies;
12. Pregnant or lactating women, and female subjects who plan to become pregnant within 1 year after cell reinfusion or male subjects whose partners plan to become pregnant within 1 year after their cell reinfusion;
13. Any unsuitable to participate in this trial judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 12 months.
  Count the Incidence of adverse events.

SECONDARY OUTCOMES:
Levels of peripheral blood γδ T cells after infusion（PK） | Up to 12 months.
  γδ T cells in the peripheral blood after infusion
Concentration of Cytokine after Infusion (PD) | Up to 12 months.
  Calculate the change in cytokine concentrations in peripheral blood after γδ T cell infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Donghua Zhang, MD, Study Director — Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology